CLINICAL TRIAL: NCT06120244
Title: Establishment of a Biobank of Nasal Epithelium Samples From Healthy Volunteers
Brief Title: Establishment of Biobank of Nasal Epithelium Samples From Healthy Volunteers
Status: Recruiting | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 10001862; 001862-I
Record Dates: First submitted 2023-11-04; First posted 2023-11-07 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07-08

CONDITIONS: Healthy
Keywords: Nasal Epithelium

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Healthy Volunteers: Healthy volunteers aged 18 years and older

SUMMARY:
Background:

Infections in the lower respiratory tract (lungs) are the leading cause of death from infectious disease worldwide. This was true even before the COVID-19 pandemic. Respiratory viruses are still a major health threat. Many of these viruses infect people by penetrating the thin skin that lines the nose. These viruses can also spread easily to other people when they multiply in the tissues that line the nose. Researchers want to learn more about what these viruses do inside the nose, how they get from the nose to the lungs, and how they spread from person to person.

Objective:

To collect cell samples from inside the noses of healthy people. These cells will be stored for use in future research on respiratory diseases.

Eligibility:

Healthy volunteers aged 18 years and older.

Design:

Most participants will have 1 visit on 1 day. They will be asked questions. Those who have a runny nose, coughing, congestion, or fever will be asked to wait up to 21 days before participating.

Participants will be given a slender swab with small bristles at the end. They will rub the inside of their nose with the swab. A clinic staff member will be present to help, if needed.

Participants will provide their name, age, and sex. This information will be encoded so that only certain researchers will know the participants identities.

Participants will not be contacted again....

DETAILED DESCRIPTION:
Study Description:

This is a repository protocol with prospective sample collection to provide samples needed for future studies of the pathogenesis of emerging respiratory viruses. Nasal brushings will be collected from approximately 100 healthy volunteers at RML and stored in the LV to be made available for future research studies that will be conducted under separate protocols, as applicable.

Primary Objective:

To obtain nasal epithelium brushes from healthy volunteers for 1) establishment of upper respiratory tract organoids, 2) assay validation, and 3) use for research into the pathogenesis of emerging respiratory viruses.

ELIGIBILITY:
* INCLUSION CRITERIA:

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

* Aged >=18 years.
* Able to provide informed consent.
* Willing to allow biological samples and data to be stored for future research.

EXCLUSION CRITERIA:

An individual who meets any of the following criteria will be excluded from participation in this

study:

* History of respiratory symptoms including but not limited to runny nose, coughing, congestion, and/or fever within the past 14 days.
* NIH and laboratory staff with direct involvement in the operation or maintenance of the repository are excluded from participation.
* An individual who has any condition that, in the judgment of the investigator, may put them at undue risk or make them unsuitable for participation in the study will be excluded.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy volunteers, aged 18 years and older, may be recruited from the general public, people working at and/or visiting Rocky Mountain Laboratories (RML), and NIH staff members and their family/contacts.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2033-10-31 (Estimated); Study Completion 2033-10-31 (Estimated)

PRIMARY OUTCOMES:
To obtain nasal epithelium brushes from healthy volunteers for 1) establishment of upper respiratory tract organoids, 2) assay validation, and 3) use for research into the pathogenesis of emerging respiratory viruses. | 10 years
  To obtain nasal epithelium brushes from healthy volunteers for 1) establishment of upper respiratory tract organoids, 2) assay validation, and 3) use for research into the pathogenesis of emerging respiratory viruses.

CONTACTS AND LOCATIONS:
Overall Officials: Emmie de Wit, Ph.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- Rocky Mountain Laboratories, Hamilton, Montana, United States

IPD SHARING:
Plan to Share IPD: Yes
IPD underlying published data will be shared upon request after appropriate collaboration agreements are in place.
Supporting Information: Study Protocol
Time Frame: At time of publication or establishment of collaboration agreement; IPD will be shared permanently.
Access Criteria: Subject level data (sex and age of donor) may be shared as part of a scientific publication. Otherwise, subject level data will be shared upon request after appropriate collaboration agreements are in place.

REFERENCES:
- [Background] Rajan A, Weaver AM, Aloisio GM, Jelinski J, Johnson HL, Venable SF, McBride T, Aideyan L, Piedra FA, Ye X, Melicoff-Portillo E, Yerramilli MRK, Zeng XL, Mancini MA, Stossi F, Maresso AW, Kotkar SA, Estes MK, Blutt S, Avadhanula V, Piedra PA. The Human Nose Organoid Respiratory Virus Model: an Ex Vivo Human Challenge Model To Study Respiratory Syncytial Virus (RSV) and Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2) Pathogenesis and Evaluate Therapeutics. mBio. 2021 Feb 22;13(1):e0351121. doi: 10.1128/mbio.03511-21. Epub 2022 Feb 15. PMID 35164569
- [Background] Stokes AB, Kieninger E, Schogler A, Kopf BS, Casaulta C, Geiser T, Regamey N, Alves MP. Comparison of three different brushing techniques to isolate and culture primary nasal epithelial cells from human subjects. Exp Lung Res. 2014 Sep;40(7):327-32. doi: 10.3109/01902148.2014.925987. Epub 2014 Jul 24. PMID 25058379